CLINICAL TRIAL: NCT05160714
Title: Individualized Response-adaptive Radiation Dose Prescription in HNC Based on MRI - Real-time ADC-guided Response Adaptive Boost in HNC - "Individuelle MR-basierte Dosisverschreibung Bei Kopf-Hals-Tumoren - ADC-basierter Adaptiver Boost"
Brief Title: Individualized Response-adaptive Radiation Dose Prescription in HNC Based on MRI
Acronym: MRL-02
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 081/2021B01
Record Dates: First submitted 2021-06-01; First posted 2021-12-16 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-03

CONDITIONS: Head and Neck Cancer
Keywords: Radiotherapy; MR-guided Radiotherapy; dose-finding study; MR-Linac; ADC-guided response adaptive Boost
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose-finding phase 1 trial with four dose levels and 3+3 design: 12 patients if no DLT occurs up to 24 patients if 1 DLT per dose-level occurs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptive SBRT Boost (Experimental): Dose-escalated SBRT boost to an ADC-based high risk subvolume in HNC
  Interventions: Radiation: Real-time ADC-guided response adaptive Boost in HNC

INTERVENTIONS:
Radiation: Real-time ADC-guided response adaptive Boost in HNC — 40 Gy in 20 fractions over 5 weeks (Monday to Thursday) to the adjuvant neck, simultaneous integrated boost with 56 Gy in 20 fractions in 5 weeks to the low-risk macroscopic tumor.
  Once weekly Dose-escalated SBRT adaptive boost to an ADC-based high risk subvolume with graduated dose levels of 5x5 Gy, 5x5.5 Gy, 5x6 Gy, 5x6.5 Gy

SUMMARY:
This Phase 1 dose-finding study investigates the maximal tolerated dose for a subsequent phase 2 trial testing MR-guided individualized response-adaptive dose prescription in HNC.

DETAILED DESCRIPTION:
This single-center, non-randomized interventional dose-finding phase I trial evaluates the maximal tolerated boost dose with respect to dose limiting toxicities in patients with locally advanced head and neck squamous cell carcinoma (UICC stage III/IVB) with an indication for a primary radiochemotherapy. The primary aim of the trial is to define the maximal tolerated dose in an ADC-based subvolume using an adaptive SBRT-boost areal. Dose-escalated SBRT boost to ADC-high risk volume will be delivered once a week and is defined according to the the actual imaging immediately performed prior to delivery (real-time adaptive) i.e. it can vary from one week to another and it might also be reduced throughout the course of treatment (response adaptive). In case of complete disappearance of high-risk subvolumes sufficient large enough to boost (<5ml), no further ADC boost but only the floor-boost dose is given. The dose escalation of the ADC-high risk volume boost is graduated in four dose levels of 5x5 Gy, 5x5.5 Gy, 5x6 Gy, 5x6.5 Gy in a classical 3+3 dose-finding design where 3 patients per radiation dose level are enrolled. Primary endpoint is the dose limiting toxicity, any acute and late non-hematologic grade 4 or 5 related to the radiotherapy intervention, ≥ grade 3 CTC v.5. oral mucositis at 3 months after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 18 years
* WHO (ECOG) performance status 0-2
* Histological proven HNC (squamous cell carcinoma)
* HPV negative tumors or high risk HPV positive tumors
* Stage III - IVB HNC of the hypopharynx, oropharynx and oral cavity according to UICC and AJCC guidelines
* Tumor extension and localization suitable for radiochemotherapy with curative intent
* Simultaneous standard chemotherapy with cisplatin applicable (no contra-indications)
* Dental examination and -treatment before start of therapy
* For women with childbearing potential and men in reproductive ages adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Refusal of the patients to take part in the trial
* Presence of distant metastases (UICC stage IVC)
* HPV positive tumors UICC Stage III with T1/2 N3, despite of smoking status
* Previous radiotherapy in the head and neck region
* Second malignancy that is likely to require treatment during the trial intervention or follow-up period or that, in the opinion of the physician, has a considerable risk of recurrence or metastases within the follow-up period
* Serious disease or medical condition with life expectancy of less than one year
* Participation in competing interventional trial on cancer treatment
* Patients who are not suitable for radiochemotherapy
* Pregnant or lactating women
* Patients not able to understand the character and individual consequences of the trial
* Nasopharyngeal and glottis laryngeal carcinomas
* Patients with contraindications for magnet-resonance tomography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | At 3 months after radiotherapy
  Dose limiting toxicity (DLT): any acute and late grade 4 or 5 related to the intervention, ≥ grade 3 CTC v.5. oral mucositis at 3 months after radiotherapy (persistent mucosal ulceration or inflammation in the high dose region with severe pain; interfering with oral intake; limiting self-care ADL)

SECONDARY OUTCOMES:
Regional tumor control | After 6 weeks, 3 months and every 3 months up to two years
  Regional tumor control will be measured by clinical H&N examinations at six weeks and then every three months up to two years. Imaging follow-up includes MRI at 6 weeks and 3 months, FDG-PET CT at 3 months and further CTs every 3 month.
Disease free survival | During treatment and after 6 weeks, 3 months and every 3 months up to two years
  Clinical H&N examinations at six weeks and then every three months up to two years, including MRI at 6 weeks and 3 months, FDG-PET CT at 3 months and further CTs every 3 month.

CONTACTS AND LOCATIONS:
Locations (1):
- UKT Radiooncology, Tübingen, Baden-Wurttemberg, Germany